CLINICAL TRIAL: NCT03476317
Title: An Open-Label Pilot Study of Fundamental Modification of the Gut Microbiota in the Treatment of Refractory Crohn's Disease
Brief Title: Pilot Study of Fundamental Modification of the Gut Microbiota in the Treatment of Refractory Crohn's Disease
Acronym: Holiday
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-014343; 5K23DK109136-02 (NIH)
Record Dates: First submitted 2018-01-08; First posted 2018-03-26 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Vancomycin; Neomycin; Ciprofloxacin; polyethylene glycol 3350; Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1-Fluconazole (Experimental): Vancomycin oral suspension four times daily (Day 1-14), plus neomycin orally three times daily (Days 1-3), plus ciprofloxacin orally twice daily (Day 4-14), plus Polyethylene Glycol 3350 (Miralax) dissolved in Gatorade on day 2, plus fluconazole orally once daily (Day 1-14).
  Interventions: Drug: Vancomycin; Drug: Neomycin; Drug: Ciprofloxacin; Drug: Polyethylene Glycol 3350; Drug: Fluconazole
- Group 1-Placebo (Placebo Comparator): Vancomycin oral suspension four times daily (Day 1-14), plus neomycin orally three times daily (Days 1-3), plus ciprofloxacin orally twice daily (Day 4-14), plus Polyethylene Glycol 3350 (Miralax) dissolved in Gatorade on day 2, plus placebo.
  Interventions: Drug: Vancomycin; Drug: Neomycin; Drug: Ciprofloxacin; Drug: Polyethylene Glycol 3350
- Group 2 (No Intervention): Collect stool samples for calprotectin in patients undergoing colonoscopy for clinical care to evaluate effect of bowel lavage alone on calprotectin.

INTERVENTIONS:
Drug: Vancomycin — Oral suspension 4 times daily (Day 1-14)
  Other Names: Vancocin
  Arms: Group 1-Fluconazole; Group 1-Placebo
Drug: Neomycin — Oral three times daily (Days 1-3)
  Other Names: Neo-Fradin
  Arms: Group 1-Fluconazole; Group 1-Placebo
Drug: Ciprofloxacin — Oral twice daily (Days 4-14)
  Other Names: Cipro
  Arms: Group 1-Fluconazole; Group 1-Placebo
Drug: Polyethylene Glycol 3350 — Dissolved in Gatorade on day 2
  Other Names: Miralax
  Arms: Group 1-Fluconazole; Group 1-Placebo
Drug: Fluconazole — Orally once daily (Day 1-14)
  Other Names: Diflucan
  Arms: Group 1-Fluconazole

SUMMARY:
The purpose of this study is to determine the effect of a novel gut microbiota-targeted therapeutic regimen (bowel lavage and antibiotics with or without an antifungal) in the management of active Crohn's Disease (CD) or indeterminate colitis (IBDU) that is refractory to conventional, immunosuppressive therapy. In addition, the study will determine the effect of PEG lavage alone on fecal calprotectin and gut microbiota in patients who are undergoing a PEG lavage for clinical care.

DETAILED DESCRIPTION:
Investigators will evaluate the efficacy of a novel treatment regimen, employing non-immunosuppressive medications, in the management of refractory CD or IBDU. Refractory patients include those patients who have experienced loss of responsiveness (LOR) or primary nonresponse to an immunomodulator or a biologic. Investigators will treat participants with a combination of gut microbiota-targeted therapies to restore a healthy gut microbiome composition. Investigators believe that this strategy will both treat the gut inflammation associated with inflammatory bowel disease (IBD) as well as salvage response to immune suppressive therapies.

Investigators will also evaluate the effect of PEG lavage alone on fecal calprotectin and gut microbiota. Participants in this arm, will be undergoing a PEG lavage in preparation for a endoscopy for clinical care. They will be asked to provide stool samples, prior to and after their PEG lavage. Participants will not be receiving any investigational treatments.

ELIGIBILITY:
Group 1

Inclusion Criteria:

* Males or females 6-18 years of age
* Current weight >10 kg (or 22 lb)
* Ability to swallow pills
* Normal kidney function
* Normal Aspartate transaminase (AST), Alanine transaminase (ALT), and alkaline phosphatase
* Active CD or IBDU defined as PCDAI ≥ 30
* C-Reactive Protein (CRP) ≥ 15mg/L (or 1.5mg/dL) or fecal calprotectin (FCP)>350mcg/g (within one month of enrollment)
* Have been treated with one of the following therapies for at least 8 weeks with primary nonresponse or an initial response, followed by loss of response [LOR] (self-reported worsening of symptoms for ≥ 7 days): azathioprine, 6-mercaptopurine, methotrexate, adalimumab, certolizumab, golimumab, infliximab, natalizumab, vedolizumab, or ustekinumab **These medications must have been administered at standard, therapeutic dosages.

Exclusion Criteria:

* Known allergy or intolerance to aminoglycosides or any of the medications used in this study
* Current use of one or more of the following medications: 5-fluorouracil, digoxin, anticoagulants, theophylline, phenytoin, probenecid, duloxetine, clozapine, sildenafil, hydrochlorothiazide, cyclosporine, hypoglycemics, terfenadine, tacrolimus, rifabutin, midazolam, and voriconazole
* Known diagnosis of diabetes mellitus
* Known or suspected structuring disease producing obstructive symptoms
* Active Clostridium difficile infection
* Prolonged QTc interval as seen on enrollment EKG
* Current use of antibiotics
* Starting or increasing the dose of an IBD related medication within 4 weeks of screening

Group 2

Inclusion Criteria

* Males or females 10 years of age and older.
* Patients undergoing a clinical GI endoscopy due to suspicion for active intestinal inflammation determined by physician global assessment (PGA).
* Undergoing a bowel preparation as part of clinical care.
* Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria

* Antibiotic use within the past 30 days.
* Current presence of an ostomy bag.
* Patients undergoing a non- polyethylene glycol 3350 cleanout.
* Unwillingness to provide informed consent.
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Albenberg, DO, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1-Fluconazole | Group 1-Placebo | Group 2
Started | 0 (Group 1 study was not completed) | 0 (Group 1 study was not completed) | 10
Completed | 0 (Group 1 study was not completed) | 0 (Group 1 study was not completed) | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: An identical study was simultaneously enrolling adult patients and results from the adult study were sufficient to make a conclusion without enrolling children. (NCT02765256)
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1-Fluconazole | Group 1-Placebo | Group 2 | Total
Number analyzed (Participants) | 0 | 0 | 10 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  |  | 9 | 9
  Between 18 and 65 years |  |  | 1 | 1
  >=65 years |  |  | 0 | 0
Age, Continuous [Median (Full Range); unit: years] |  |  | 16.5 [11 to 20] | 16.5 [11 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 2 | 2
  Male |  |  | 8 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States |  |  | 10 | 10
Calprotectin [Median (Full Range); unit: mcg/g] |  |  | 1254.5 [511 to 3000] | 1254.5 [511 to 3000]

OUTCOME MEASURES:

1. Primary Outcome: Change in FCP in Group 2 Participants
Description: Change in fecal calprotectin between stool samples collected at baseline and day 12 after procedure in Group 2 participants.
Time Frame: change from baseline to day 12
Population: Group 1 study was not done.
Measure: Median (Full Range); unit: mcg/g
Arm/Group | Group 1-Fluconazole | Group 1-Placebo | Group 2
Number analyzed (Participants) | 0 | 0 | 10
mcg/g |  |  | 1501 [271 to 3000]
Statistical Analysis 1: Comparison: Group 2; Test type: Equivalence — Median difference in calprotectin for controls from day 12 to baseline; p = 1.0, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Disease Activity by Pediatric Crohn's Disease Activity Index
Description: The primary endpoint will be the change in disease activity, as measured by Pediatric Crohn's Disease Activity Index (PCDAI) score, between the enrollment visit and Day 15. All participants who withdraw for any reason prior to day 15 will be considered treatment failures. The Pediatric Crohn's Disease Activity Index is a clinical score which takes into account general well being, degree of abdominal pain, number of liquid stools per day, abdominal physical examination, and Crohn's disease complications.
Time Frame: Baseline, Day 15
Population: This outcome was specific to Group 1 and we did not enroll patients into Group1as an identical study was simultaneously enrolling adult patients and results from the adult study were sufficient to make a conclusion without enrolling children.
Arm/Group | Group 1-Fluconazole | Group 1-Placebo | Group 2
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Change in Disease Activity by Fecal Calprotectin (FCP)
Description: The second primary outcome measure will be the change in disease activity, as measured by fecal calprotectin, between the enrollment visit and day 15. The fecal calprotectin is a stool test which measures intestinal inflammation.
Time Frame: Baseline, Day 15
Population: This outcome was specific to Group 1 and Group 1 study was not completed.
Arm/Group | Group 1-Fluconazole | Group 1-Placebo | Group 2
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change in C-reactive Protein (CRP)
Description: A secondary outcome measure will be the change in C-reactive protein between the enrollment visit and day 15. The C-reactive protein is a blood test which measures systemic inflammation.
Time Frame: Baseline, Day 15
Population: This outcome was specific to Group 1 and Group 1 study was not completed.
Arm/Group | Group 1-Fluconazole | Group 1-Placebo | Group 2
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Safety and Tolerability of the Treatment Regimen Based on Medication Side Effects and/or Adverse Events
Time Frame: 105 days
Population: This outcome is specific to Group 1 and Group 1 study was not completed.
Arm/Group | Group 1-Fluconazole | Group 1-Placebo | Group 2
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 days
Description: Group 1 study was not completed
Arm/Group | Group 1-Fluconazole | Group 1-Placebo | Group 2
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/10
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/10

LIMITATIONS AND CAVEATS:
Group 1 study was not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT03476317/Prot_SAP_001.pdf
  • Informed Consent Form (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT03476317/ICF_000.pdf